CLINICAL TRIAL: NCT05627063
Title: A Phase 1, Open-Label Study of ABSK121-NX to Assess Safety, Tolerability, and Pharmacokinetics in Patients With Advanced Solid Tumors
Brief Title: A Study to Assess Safety, Tolerability, and Pharmacokinetics of ABSK121-NX in Patients With Advanced Solid Tumors
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Abbisko Therapeutics Co, Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ABSK121-NX-101
Record Dates: First submitted 2022-11-15; First posted 2022-11-25 (Actual); Last update posted 2025-10-20 (Actual); Status verified 2025-10

CONDITIONS: Solid Tumor

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- ABSK121-NX (Experimental): Dose escalation of oral ABSK121-NX will be guided by the Bayesian optimal interval (BOIN) design based on safety data collected until a maximum tolerated dose (MTD) or maximum administered dose (MAD) has been identified. Patients will receive a single dose of ABSK121-NX on Day -7 followed by a 7-day washout, as a run-in period to access the safety and PK of ABSK121-NX. Then, patients will continuously receive ABSK121-NX once daily (QD).
  The dose escalation will start at 3 mg QD followed by dose escalation of a total of 8 potential dose levels. Once RDE is determined, an RDE-confirmation group of up to 24 more patients may be enrolled at the selected dose levels to further evaluate safety and efficacy (up to 12 per dose level/regimen), if approved by the sponsor. In addition, a preliminary food-effect (FE) may be evaluated in at least 6 patients from the RDE- confirmation part.
  After the RDE is confirmed in the dose Escalation part, the dose Expansion phase will be conducted.
  Interventions: Drug: ABSK121-NX

INTERVENTIONS:
Drug: ABSK121-NX — In the escalation part, patients will receive a single dose of oral ABSK121-NX on Day -7 followed by a 7-day washout (Day -7 dosing day as 1st day of wash out) as a run-in period to access the safety and PK of ABSK121-NX. Then, patients will continuously receive ABSK121-NX once daily (QD) starting at C1D1 and continuing in subsequent cycles (28-day cycles). The starting dose is 3mg QD. In the expansion part, patients will each receive oral ABSK121-NX at the RDE in repeated 28-day cycles.

SUMMARY:
This is an open-label phase 1 study with expansion. The study will start with a dose escalation of single-agent ABSK121-NX administered in repeated 28-day cycles in patients with advanced solid tumors to evaluate safety and tolerability. The expansion part will investigate oral ABSK121-NX at the recommended dose for expansion (RDE) to further evaluate safety and tolerability among selected tumor types. Preliminary antitumor activity will also be assessed.

DETAILED DESCRIPTION:
Escalation Part:

Dose escalation of oral ABSK121-NX will be guided by the Bayesian optimal interval (BOIN) design based on safety data collected until a maximum tolerated dose (MTD) or maximum administered dose (MAD) has been identified. During the dose escalation part of the study, patients will receive a single dose of ABSK121 on Day -7 followed by a 7-day washout (Day -7 dosing day as 1st day of wash out) as a run-in period to access the safety and PK of ABSK121-NX. Then, patients will continuously receive ABSK121-NX once daily (QD) beginning at C1D1.

The dose escalation will start at 3 mg QD followed by dose escalation of a total of 8 potential dose levels. Once RDE is determined, an RDE-confirmation group of up to 24 more patients may be enrolled at the selected dose levels to further evaluate safety and efficacy (up to 12 per dose level/regimen), if approved by the sponsor. In addition, a preliminary food-effect (FE) may be evaluated in Cycle 1 D15 or later in at least 6 patients from the RDE- confirmation part.

After the RDE is determined in the dose escalation part, the dose expansion phase will be conducted.

Expansion Part:

When health authorities outside US require that the safety data in the local population be provided prior to the expansion part, a minimum of 3 local subjects will be enrolled and treated at the selected RDE dose level first in that country/region to evaluate the tolerability of ABSK121-NX. The inclusion and exclusion criteria for escalation part will apply for these subjects. After similar safety and tolerability of ABSK121-NX in patients in the relevant locality have been confirmed by local Investigators and the Sponsor, additional patients will be allowed to enroll in the expansion part.

ELIGIBILITY:
Inclusion Criteria:

1. Patients should understand, sign, and date the written informed consent form prior to screening
2. Male or female age 18 years or older
3. Patients with histologically confirmed locally-advanced or metastatic solid tumors who have progressed on, or are intolerant of standard therapy, or for whom no standard therapy exists, or reject standard therapy

For RDE-confirmation in the escalation part: patients with selected advanced solid tumors, i.e.,

1. Patients must have the following FGFR genetic alterations based on central laboratory tests or existing test reports of tumor tissue and/or blood:

   1. Urothelial carcinoma (UC): pre-specified FGFR3 mutations (R248C, S249C, G370C, Y373C) or FGFR2/3 fusions (partner gene is previously described or in frame), or
   2. Intrahepatic Cholangiocarcinoma (iCCA): FGFR2 fusions or rearrangements which containing an intact kinase domain as follows:

      • FGFR2 fusions: FGFR2 rearrangements with a literature-derived known partner gene regardless of strand or frame, or FGFR2 rearrangements in the same 5' to 3' orientation and in frame with a novel partner gene

      • FGFR2 rearrangements: FGFR2 rearrangements with one breakpoint in the hotspot region (intron 17-exon 18) and the other breakpoint in an intergenic region or within another gene, or intragenic duplication of the kinase domain (exon 9-17)
2. Patients must have at least one measurable target lesion according to RECIST 1.1

For the expansion Part:

1) Patients must have the following FGFR genetic alterations based on central laboratory tests or existing test reports of tumor tissue and/or blood:

1. Urothelial carcinoma: pre-specified FGFR3 mutations (R248C, S249C, G370C, Y373C) or FGFR2/3 fusions (partner gene is previously described or in frame)
2. Cholangiocarcinoma: FGFR2 fusions or rearrangements which containing an intact kinase domain as follows:

   * FGFR2 fusions: FGFR2 rearrangements with a literature-derived known partner gene regardless of strand or frame, or FGFR2 rearrangements in the same 5' to 3' orientation and in frame with a novel partner gene
   * FGFR2 rearrangements: FGFR2 rearrangements with one breakpoint in the hotspot region (intron 17-exon 18) and the other breakpoint in an intergenic region or within another gene, or intragenic duplication of the kinase domain (exon 9-17)
3. Other tumor types: solid tumors harboring FGFR1-4 alterations including activating mutations, fusions or rearrangements and amplifications, e.g., advanced/metastatic gastric cancer (GC) or gastroesophageal junction (GEJ) carcinoma harboring the FGFR2 amplifications, or iCCA patients or UC patients with other FGFR alterations not mentioned above, are also allowed

   2) Patients must have at least one measurable target lesion according to RECIST 1.1

   3) Previous FGFR inhibitors treated and progressed cohort in UC or iCCA patients: received treatment with FGFR inhibitors and experienced disease progression/recurrence during or after FGFR inhibitors treatment

   4. ECOG performance status 0 or 1

   5. Life expectancy ≥3 months

   6. Adequate organ function and bone marrow function as indicated by the following screening assessments performed within 14 days prior to the first dose of study drug:
   1. Absolute neutrophil count (ANC) ≥1.5×109/L (without the use of hematopoietic colony-stimulating growth factors (e.g. G-CSF, GM-CSF, M-CSF) within 7 days before testing)
   2. Platelet count (PLT) ≥100×109/L (without transfusion within 14 days before testing)
   3. Hemoglobin (Hb) ≥90 g/L (without transfusion within 7 days before testing)
   4. Total bilirubin (TBIL) ≤1×ULN
   5. Aspartate transaminase (AST) and alanine transaminase (ALT) ≤2.5×ULN
   6. Creatinine clearance (Crcl) ≥60 mL/min based on Cockcroft-Gault formula
   7. Electrolyte: magnesium within 0.85 to 1.25 × institutional normal limits, sodium ≥130 mmol/L, potassium within institutional normal limits 7. For patients participating exploration of food effect:

   <!-- -->

   1. be able to eat a standardized high-fat, high caloric meal within 30 minutes
   2. be able to fast for 10 hours

   Exclusion Criteria:
   1. Known allergy or hypersensitivity to any component of the investigational product
   2. RDE-confirmation in Escalation part: Prior treatment with any FGFR inhibitors
   3. Expansion part:

   <!-- -->

   1. Previously FGFR-inhibitors naive cohorts in UC or iCCA patients: Prior treatment with any FGFR inhibitors
   2. Other solid tumors cohort: Prior treatment with any FGFR inhibitors

   4. Has a known additional malignancy that is progressing or has required active treatment.

   5. Has persistent phosphate level >ULN during screening (within 14 days prior to the first dose of study treatment) and despite medical management

   6. Unable to swallow capsules or tablets or malabsorption syndrome, disease significantly affecting GI function, or resection of the stomach or small bowel, symptomatic inflammatory bowel disease or ulcerative colitis, or partial or complete bowel obstruction. If any of these conditions exist, the site should discuss with the sponsor to determine patient eligibility

   7. Previous anti-cancer therapy, including chemotherapy (chemotherapy with nitrosourea or mitomycin received ≤ 6 weeks prior to initiation of study treatment), radiotherapy, molecular targeted therapy, antibody therapy or other investigational drugs received ≤4 weeks; endocrine therapy ≤2 weeks or ≤5 half-lives (whichever is shorter) prior to initiation of study treatment

   8. Major surgery within 4 weeks of the first dose of study drug. Note that all surgical wounds must be healed and free of infection or dehiscence

   9. Prior toxicities from chemotherapy, radiotherapy, and other anti-cancer therapies, including immunotherapy that have not regressed to Grade ≤1 severity (CTCAE v5.0) with the exception of alopecia, vitiligo and grade 2 peripheral neurotoxicity

   10. Potent inhibitors or inducers of CYP3A4 within 2 weeks before the first dose of study treatment (3 weeks for St John's Wort). Refer to https://www.fda.gov/drugs/drug-interactions-labeling/drug-development-and-drug-interactions-table-substrates-inhibitors-and-inducers for a list of drugs

   11. Active central nervous system (CNS) metastases including presence of cerebral edema, requirement for systemic steroid treatment, disease progression due to intracranial lesions, leptomeningeal metastasis, and other clinical symptoms related to CNS metastases

   12. Impaired cardiac function or clinically significant cardiac disease, including any one of the following:
   1. New York Heart Association class III or IV heart disease, active ischemia or any other uncontrolled cardiac condition such as angina pectoris, clinically significant cardiac arrhythmia requiring therapy, uncontrolled hypertension or congestive heart failure,
   2. Baseline prolongation of the rate-corrected QT interval based on repeated demonstration of QTcF >470 ms (average of screening triplicates) or history of long QT interval corrected (QTc) syndrome (Note: QTc interval corrected by Fridericia's formula),
   3. Left ventricular ejection fraction (LVEF) <50% or below the institutional lower limit of normal (whichever is higher)

   13. Known acquired immunodeficiency syndrome (AIDS)-related illness, or positive test for HIV 1/2 antibody

   14. Exclusion of hepatitis infection based on the following results and/or criteria:
   1. Active hepatitis B infection: positive tests for hepatitis B surface antigen (HBsAg), or antibody to hepatitis B core antigen (anti-HBc). A patient with positive tests for HBsAg or anti-HBc but with HBV-DNA measurements lower than detectable (or per local practice) can be enrolled,
   2. Active hepatitis C infection: positive Hepatitis C virus antibody. If positive antibody to hepatitis C Virus (anti-HCV) is detected, Hepatitis C virus RNA by polymerase chain reaction (PCR) is necessary. A patient with positive anti-HCV but with a negative test for HCV RNA can be enrolled

   15. Any of the following ophthalmological criteria:
   1. Current evidence or previous history of retinal pigment epithelial detachment (RPED) /Central serous retinopathy (CSR)
   2. Previous laser treatment or intra-ocular injection for treatment of macular degeneration
   3. Current evidence or previous history of dry or wet age-related macular degeneration
   4. Current evidence or previous history of retinal vein occlusion (RVO)
   5. Current evidence or previous history of retinal degenerative diseases (e.g., hereditary)
   6. Diabetic retinopathy with macular edema
   7. Current evidence or previous history of any other clinically relevant chorioretinal defect
   8. Uncontrolled glaucoma or intraocular pressure > 21 mmHg [after intervention per local standard of care (SOC)]
   9. History of systemic disease or ophthalmologic disorders requiring chronic use of ophthalmic steroids
   10. Evidence of any ongoing ophthalmologic abnormalities or symptoms that are acute (within 4 weeks prior to first dose) or actively progressing
   11. Current evidence or previous history of corneal pathology such as keratopathy, corneal abrasion or ulceration, or current evidence of conjunctivitis

   16. Patients with refractory/uncontrolled ascites or pleural effusion

   17. Pregnant or nursing (lactating) women, where pregnancy is defined as the state of a female after conception and until the termination of gestation, confirmed by a positive human chorionic gonadotropin (hCG) laboratory test within 7 days prior to the start of study drug

   18. Non-surgically sterilized male or female patients of childbearing potential must agree to use highly effective methods of birth control during the study and for approximately 6 months after the last dose of study drug. A condom is also required to be used by vasectomized men to prevent delivery of the drug via seminal fluid

   19. Vaccination with a live, attenuated vaccine within 4 weeks prior to the first dose of study treatment except for administration of inactivate vaccines (e.g., COVID-19 vaccines, inactivated influenza vaccines)

   20. Any other clinically significant comorbidities, such as uncontrolled pulmonary disease, active infection, or any other condition, which in the judgment of the Investigator, could compromise compliance with the protocol, interfere with the interpretation of study results, or predispose the patient to safety risks

   21. Planned major surgery during study treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 169 (Estimated)
Dates: Start 2023-06-26 (Actual); Primary Completion 2026-03-15 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of DLT | At the end of Cycle 1 (each cycle is 28 days)
  dose-limiting toxicities (DLTs)
Incidence and severity of adverse events (AEs) | Through study completion, an average of half year
  adverse events (AEs), adverse events of special interest (AESIs) and serious adverse events (SAEs)

SECONDARY OUTCOMES:
Cmax | Through the study completion, an average of half year
  maximum observed concentration
Tmax | Through the study completion, an average of half year
  time to maximum observed concentration
AUC | Through the study completion, an average of half year
  area under the concentration-time curve
t1/2 | Through the study completion, an average of half year
  half-life
Vz/F | Through the study completion, an average of half year
  apparent volume of distribution
CL/F | Through the study completion, an average of half year
  apparent oral clearance
Cmax,ss | Through the study completion, an average of half year
  maximum observed concentration of steady/state
Cmin,ss | Through the study completion, an average of half year
  minimum observed concentration of steady/state
AUCtau,ss | Through the study completion, an average of half year
  area under the concentration-time curve after multiple dose
AR | Through the study completion, an average of half year
  accumulation ratio
ORR | Through the study completion, an average of half year
  overall response rate
DoR | Through the study completion, an average of half year
  duration of response
DCR | Through the study completion, an average of half year
  disease control rate
PFS | Through the study completion, an average of half year
  Progression-free survival
OS | Through the study completion, an average of half year
  overall survival

CONTACTS AND LOCATIONS:
Overall Officials: Yuan Lu, Study Director — Wuxi Abbisko Biomedical Technology Co., Ltd.
Locations (24):
- United States (4):
  - UC San Diego Moores Cancer Center, La Jolla, California
  - Karmanos Cancer Institute, Detroit, Michigan
  - Comprehensive Cancer Centers of Nevada, Las Vegas, Nevada
  - Gabrail Cancer Center Research, Canton, Ohio
- China (20):
  - Chongqing University Cancer Hospital, Chongqing, Chongqing Municipality
  - The First Affiliated Hospital of Henan University of Science & Technology, Luoyang, Henan
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - Hubei Cancer Hospital, Wuhan, Hubei
  - Hunan Central Hospital, Changsha, Hunan
  - The Affiliated Hospital of Inner Mongolia Medical University, Hohhot, Inner Mongolia
  - The First Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - Jilin Cancer Hospital, Changchun, Jilin
  - The First Hospital of China Medical University, Shenyang, Liaoning
  - Shanghai East Hospital Tongji University, Shanghai, Shanghai Municipality
  - Shanxi Provincial Cancer Hospital, Taiyuan, Shanxi
  - West China School of Medicine/West China Hospital of Sichuan University, Chengdu, Sichuan
  - Mianyang Central Hospital, Mianyang, Sichuan
  - Zhejiang University Cancer Hospital, Hangzhou, Zhejiang
  - Fujian Cancer Hospital (Department of Hepatobiliary and Pancreatic Oncology /Phase I Ward), Fuzhou
  - Harbin Medical University Cancer Hospital (Gastroenterology Department 2nd Ward), Haerbin
  - Zhongshan Hospital of Fudan University (Hepatological Surgery Department), Shanghai
  - Zhongshan Hospital of Fudan University (Medical Oncology Department), Shanghai
  - Liaoning Cancer Hospital (Phase I Ward), Shenyang
  - Yantai Yuhuangding Hospital (Department of Medical Oncology, 1), Yantai

IPD SHARING:
Plan to Share IPD: No